CLINICAL TRIAL: NCT05272306
Title: The Utility of Gastro-laryngeal Tube During Transesophageal Echocardiography: Prospective Randomized Clinical Trial
Brief Title: Gastro-laryngeal Tube During Transesophageal Echocardiography
Acronym: GLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muhittin Calim, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: muhittincalim1
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia; Sedation; Analgesia; Airway Complication of Anesthesia
Keywords: Anesthesia; Sedation; Analgesia; Gastro-laryngeal tube; Transesophageal echocardiography
MeSH Terms: conditions — Agnosia | interventions — Pain Measurement

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation and Analgesia (Active Comparator): A standardized sedation and analgesia will be administered by an experienced anesthesiologist. After administration of lidocaine and atropine sulfate, and also preoxygenation (100% 4 L/min oxygen for 3 minutes), patients will be induced with propofol and fentanyl via intravenous route at doses calculated according to ideal body weight. Anesthesia was maintained with propofol infusion. Repetitive intravenous boluses of propofol will be administered, if required. Patients will be received oxygen (100%, 3 L/min) through a nasal cannula during sedation and analgesia.
  Interventions: Other: Number of attempts for successful transesophageal echocardiography; Diagnostic Test: A questionnaire for cardiologist satisfaction; Diagnostic Test: A questionnaire for patient satisfaction
- Gastro-laryngeal Tube (Active Comparator): After administration of lidocaine and atropine sulfate, and also preoxygenation (100% 4 L/min oxygen for 3 min), patients will be induced with propofol and fentanyl. After induction of anesthesia, supraglottic airway device named Gastro-laryngeal Tube (GLT) will be inserted. Patients will be ventilated mechanically with a tidal volume of 6-8 mL/kg based on ideal body weight and a frequency of 12-14 breaths/min after inserting the GLT. Repetitive intravenous boluses of propofol will be administered, if required.
  Interventions: Other: Number of attempts for successful transesophageal echocardiography; Diagnostic Test: A questionnaire for cardiologist satisfaction; Diagnostic Test: A questionnaire for patient satisfaction

INTERVENTIONS:
Other: Number of attempts for successful transesophageal echocardiography — Transesophageal echocardiography probe will be inserted after induction of anesthesia. Number of attempts for successful transesophageal echocardiography will be recorded.
  Other Names: TEE
Diagnostic Test: A questionnaire for cardiologist satisfaction — A questionnaire for cardiologist satisfaction will be measured on a grade of 0-4 (1= very bad, 2= bad, 3= good, 4= very good).
  Other Names: Questionnaire
Diagnostic Test: A questionnaire for patient satisfaction — A questionnaire for patient satisfaction will be measured on a grade of 0-4 (1= very bad, 2= bad, 3= good, 4= very good).
  Other Names: Questionnaire

SUMMARY:
To analyze the effects of the use of Gastro-laryngeal Tube on intraoperative and postoperative hemodynamics, procedure comfort, and cardiologist and patient satisfactions during transesophageal echocardiography.

DETAILED DESCRIPTION:
Transesophageal echocardiography (TEE) is an ultrasonic imaging method providing anatomic, functional and hemodynamic information by imaging the heart and thoracic vascular structures using a probe advanced through the esophagus toward the stomach. The probe, with an ultrasonic wave converter at the tip, is placed in the patient's esophagus and begins assessment at the closest location to the heart. This position allows detailed assessment of the heart. It is commonly used during heart surgery, while it is also used in outpatient practice during cardiology examinations for diagnostic purposes.

Currently, TEE is performed with the outpatient admission concept in procedure rooms of the relevant departments as a semi-invasive procedure. TEE provides relatively higher quality and detailed assessments compared to transthoracic echocardiography (TTE). When images obtained with TEE are compared with TTE images, posterior structures like the interatrial septum, mitral valve, left atrium and pulmonary veins were reported to be assessed at superior levels. In addition to this advantage of TEE, the presence of the TEE probe in the oropharyngeal passage and need for deep sedation involve high complication risks. During sedation administration, the common use of the oropharyngeal passage by both cardiologist and anesthesiologist forms a risk in terms of airway management. Especially during deep sedation and analgesia, special equipment and manipulation may be required for the safety of airway management.

In modern medical approaches, priority has begun to be given to procedure comfort, along with diagnosis and treatment of the patient. With this aim, endoscopic esophagus procedures are frequently performed under sedation. Sedation administration is not an innocent procedure, and management includes many difficulties. The incidence of complications related anesthesia and the procedure is variable, but hypoxia, unplanned endotracheal intubation secondary to desaturation or aspiration, accidental tracheal insertion of gastroscope, bronchospasm, laryngospasm and hemodynamic instability may be encountered. A review of the literature stated the hypoxia incidence related to sedation was 1.5-70%. The broad interval of incidence is stated to be linked to the use, or not, of airway protective approaches.

The importance given to patient comfort and satisfaction and desire of endoscopist to perform procedures more reliably and with shared responsibility have opened the door to new research and innovations. This demand has motivated industry to develop new pharmaceutical agents and medical instruments. The gastro-laryngeal tube (GLT) is designed with the aim of ensuring the safety of airway management and optimum performance of endoscopy for esophageal procedures under deep sedation and is a new tool offered for use. GLT is a modification of a laryngeal tube allowing passage of the gastroscope or TEE probe, a suitable channel for manipulation and ensuring supraglottic airway control at the same time. There are two inflatable cuffs, one within the esophagus and the other in the hypopharynx. These cuffs ensure airway safety and stabilization of the gastro-laryngeal tube.

The investigators hypothesized that GLT, allowing passage of the TEE probe and ensuring supraglottic airway control, would provide more advantages in terms of hemodynamic stabilization, complications related airway management, cardiologist and patient satisfactions when used in a clinical setting. To date, there has been no detailed prospective clinical study analyzing the performance of the GLT during TEE. The present study sought to address this gap by performing a prospective clinical study to analyze the performance of the GLT during TEE. Primary outcome measures were safety of airway management, and cardiologist and patient satisfactions. This study also recorded demographic characteristics, intraoperative and postoperative hemodynamics, level of hypoxemia, and duration of procedure as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-II
* Aged 20-75 years old

Exclusion Criteria:

* Under 20 years old
* Over 75 years old
* An allergy to anesthetic drugs
* Emergent procedure
* Uncontrolled cerebrovascular disease
* Drug and alcohol addiction
* Performed oropharyngeal surgery
* Patients who refused written informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
A questionnaire for cardiologist satisfaction | A questionnaire will be performed to cardiologist 30 minutes after the procedure
  A questionnaire for cardiologist satisfaction will be measured on a grade of 0-4 (1= very bad, 2= bad, 3= good, 4= very good).

SECONDARY OUTCOMES:
Number of attempts for successful transesophageal echocardiography | Transesophageal echocardiography probe will be inserted during the procedure.
  Transesophageal echocardiography probe will be inserted after induction of anesthesia. Number of attempts for successful transesophageal echocardiography will be recorded.
A questionnaire for patient satisfaction | A questionnaire will be performed to the all patients 2 hours after the procedure
  A questionnaire for patient satisfaction will be measured on a grade of 0-4 (1= very bad, 2= bad, 3= good, 4= very good).
Heart rate | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Heart rate is measured as beats/minute on the anesthesia monitor
Mean arterial pressure | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Mean arterial pressure is measured as mmHg on the anesthesia monitor
Peripheral oxygen saturation | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Peripheral oxygen saturation is measured as percentage (%) on the anesthesia monitor

CONTACTS AND LOCATIONS:
Overall Officials: Muhittin Calim, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Muhittin Calim, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daskaya H, Uysal H, Ciftci T, Baysal B, Idin K, Karaaslan K. Use of the gastro-laryngeal tube in endoscopic retrograde cholangiopancreatography cases under sedation/analgesia. Turk J Gastroenterol. 2016 May;27(3):246-51. doi: 10.5152/tjg.2016.16121. PMID 27210780

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT05272306/Prot_SAP_001.pdf